CLINICAL TRIAL: NCT03770234
Title: Investigation of the Pharmacokinetics of a Transtec® 35 µg/h Transdermal Patch Application for 96 Hours and a Patch Application for 72 Hours in an Open, Randomised, Single Application, Two-period Crossover, Phase I Study in 30 Healthy Male Volunteers
Brief Title: Clinical Study in Healthy Men to Investigate the Uptake of Buprenorphine and Its Elimination From the Body After Dermal Application as Patches for 96 Hours and for 72 Hours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP5303/04
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Pain; Pharmacokinetics
MeSH Terms: conditions — Pain | interventions — Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Each participant will apply Transtec 35 µg/hour transdermal patch, once for 96 hours (Treatment A) and once for 72 hours (Treatment B) in randomized order. Between removal of the first patch and application of the second patch, there will be a washout period of at least 10 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A: Transtec patch application for 96 hours (Experimental): Transtec 35 µg/hour transdermal patch wearing period of 96 hours, with application of patch on Study Day 1 and removal on Study Day 5.
  Interventions: Drug: Transtec 35 µg/hour transdermal patch
- Treatment B: Transtec patch application for 72 hours (Experimental): Transtec 35 µg/hour transdermal patch wearing period of 72 hours, with application of patch on Study Day 1 and removal on Study Day 4.
  Interventions: Drug: Transtec 35 µg/hour transdermal patch

INTERVENTIONS:
Drug: Transtec 35 µg/hour transdermal patch — Transdermal patch containing 20 mg buprenorphine in an active surface area of 25 squared centimeters. Buprenorphine release rate 35 µg/hour.

SUMMARY:
The purpose of the study was to investigate the pharmacokinetics (i.e. the uptake, distribution and elimination from the body) of dermally applied buprenorphine during and after different application periods, i.e., a 96-hour and a 72-hour application of the Transtec (Registered Trademark) patch (release rate 35 micrograms per hour [µg/hour]). In the Transtec summary of product characteristics (prescribing information for the physician), the wearing time per patch is restricted to three days (72 hours) after which the patch has to be replaced. However, market experience has shown that the Transtec patches are sometimes worn for a period longer than three days, i.e. they sometimes happen to be only replaced every four days. There was currently no data available as how to evaluate this longer wearing period.

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasian volunteers, aged 25-45 years.
* Body mass index (BMI) between 18 and 30 kilogram/squared meter (extremes included).
* Good physical and mental health status (no current acute illness) determined on the basis of the medical history and a general clinical examination.
* Systolic blood pressure between 90 millimeter mercury (mmHg) and 150 mmHg (extremes included).
* Diastolic blood pressure between 45 mmHg and 90 mmHg (extremes included).
* Pulse rate between 45 beats per minute (bpm) and 100 bpm (extremes included).
* Electrocardiogram (12 lead) considered as normal by the investigator.
* Results of laboratory tests within the normal ranges for the testing laboratory. The investigator may include a participant having values outside the accepted range if, in his/her opinion, these values are of no clinical relevance. The decision will be justified.
* The participant has been informed using the informed consent approved by the local ethics committee.
* The consent was obtained by participant's signature.

Exclusion Criteria:

* Diseases and functional disorders of the central nervous system (CNS), endocrinological system, gastrointestinal tract, hepatobiliary system, renal system, respiratory system or cardiovascular system including marked repolarization abnormality (e.g. suspicious or definite congenital long QT syndrome) or co-medication that is known to influence cardiac repolarization substantially.
* History of seizures or at risk (i.e. head trauma, epilepsy in family anamnesis, unclear loss of consciousness).
* Malignancy.
* History of orthostatic hypotension.
* Positive human immunodeficiency virus (HIV) 1/2-antibodies, hepatitis B surface (HBs) -antigen, hepatitis B core (HBc) -antibodies, hepatitis C virus (HCV) -antibody tests at the screening examination.
* Drug allergy.
* Bronchial asthma.
* Participation in another clinical study within three month prior to the start of this study (exception: characterization of metabolizer status).
* Blood donation (more than 100 milliliters) within three month prior to the start of this study.
* Use of any medication within four weeks prior to the start of the study (self-medication or prescription).
* Evidence of alcohol, medication or drug abuse.
* Positive Naloxone challenge test.
* Positive drug abuse screening test.
* Extremely unbalanced diet (in the opinion of the investigator).
* Excessive consumption of food or beverages containing caffeine or other xanthines (more than five cups of coffee or equivalent per day).
* Smoking of more than 20 cigarettes per day.
* Neurotic personality, psychiatric illness or suicide risk.
* Known or suspected of not being able to comply with the study protocol.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-04-05 (Actual); Primary Completion 2004-05-26 (Actual); Study Completion 2004-05-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: AUC48-72 for buprenorphine | From 48 hours to 72 hours
  Partial area under the plasma concentration-time curve (from 48 hours after application until 72 hours after application).
Pharmacokinetic parameter: AUC72-96 for buprenorphine | From 72 hours to 96 hours
  Partial area under the plasma concentration-time curve (from 72 hours after application until 96 hours after application).

SECONDARY OUTCOMES:
Pharmacokinetic parameter: Cmax for buprenorphine | Before application and after 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104,112,120,132,144,156, and 168 hours
  Maximum observed plasma concentration of the measured concentration-time profile. Blood samples will be taken for the determination of buprenorphine plasma concentrations at distinct time points: Before application to 144 hours after patch application. If the patch was applied for 96 hours, additional samples were taken at 156 and 168 hours after application. For the analysis of buprenorphine in human plasma, a validated liquid chromatography mass spectrometry (LC/MS/MS)-method will be used.
Pharmacokinetic parameter: tmax for buprenorphine | Before application and after 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104,112,120,132,144,156, and 168 hours
  Time of maximum concentration, time after transdermal patch application at which Cmax occurs.
Pharmacokinetic parameter: AUC0-t for buprenorphine | Before application and after 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104,112,120,132,144,156, and 168 hours
  Area under plasma concentration-time curve from application until the last sampling point (t) with a quantifiable concentration, calculated by the linear/log trapezoidal method, i.e., the linear trapezoidal rule is applied up to Cmax and then the log trapezoidal rule is applied for the remainder of the curve.
Pharmacokinetic parameter: t1/2z for buprenorphine | Before application and after 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104,112,120,132,144,156, and 168 hours
  Apparent terminal elimination half-life.
Pharmacokinetic parameter: AUC0-inf for buprenorphine | Before application and after 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104,112,120,132,144,156, and 168 hours
  Area under the plasma concentration-time curve extrapolated to infinity.
Incidence of treatment emergent adverse events | From patch application (Day 1) until Final check (Day 12)
  Number of adverse events and number of participants with adverse events.
Characteristics of treatment emergent adverse events | From patch application (Day 1) until Final check (Day 12)
  Adverse events with information on intensity, seriousness, relationship to the investigational product, outcome and action taken will be determined.
Onset and duration of treatment emergent adverse events | From patch application (Day 1) until Final check (Day 12)
  Adverse events with information on onset and duration to the investigational product will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Institut für Klinische Pharmakologie Bobenheim, Grünstadt, Germany

IPD SHARING:
Plan to Share IPD: No